CLINICAL TRIAL: NCT06540833
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Flexible-dose Study to Assess the Efficacy, Safety, and Tolerability of ITI-1284 in Patients With Psychosis Associated With Alzheimer's Disease
Brief Title: A Study to Assess the Efficacy and Safety of ITI-1284 in the Treatment of Psychosis Associated With Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-1284-201
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Psychosis Associated With Alzheimer's Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ITI-1284 (Experimental)
  Interventions: Drug: ITI-1284
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-1284 — ITI-1284 10 mg or 20 mg rapidly disintegrating tablet, taken once daily, sublingual administration
  Arms: ITI-1284
Drug: Placebo — Placebo rapidly disintegrating tablet, taken once daily, sublingual administration
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled, flexible-dose study evaluating the efficacy, safety, and tolerability of ITI-1284 compared with placebo in the treatment of psychosis in patients with AD.

DETAILED DESCRIPTION:
The study will be conducted in 3 periods:

* Screening Period (up to 4 weeks) during which patient eligibility will be assessed;
* Double-blind Treatment Period (6 weeks) during which all patients will be randomized in a 1:1 ratio to receive either ITI-1284 or placebo;
* Safety Follow-up Period (30 days) during which all patients will return for a safety follow-up visit approximately 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Can understand the nature of the trial and protocol requirements and provide signed informed consent, if in the judgement of the Investigator is deemed competent to provide consent or if patient is deemed not competent to provide informed consent, with the patient's assent (if capable), consent may be provided by an appropriate person (eg, patient's Legally Authorized Representative [LAR]) before the initiation of any study-specific procedures in accordance with local regulations;
2. Meets clinical criteria for AD based on 2011 NIA-AA criteria and either:

   1. Has a high likelihood for amyloid pathology consistent with AD, as confirmed by blood-based biomarker at Screening; or
   2. Has documented confirmation of AD by cerebrospinal fluid (CSF) biomarker or amyloid positron emission tomography (PET) brain scan;
3. Meets criteria for psychosis in accordance with the International Psychogeriatric Association (IPA) provisional consensus definition at Screening and Baseline;
4. Scoring ≥ 2 on any item of the BEHAVE-AD Part A. Paranoid and Delusional Ideation item and/or Part B. Hallucinations item (ie, psychosis subscale) at Screening and Baseline;
5. CGI-S score ≥ 4 at Screening and Baseline;
6. Mini-Mental State Examination, 2nd Edition™: Standard Version (MMSE-2®:SV) score of 6 to 24 (inclusive) at Screening with sufficient verbal ability to understand and answer questions and comply with procedures;
7. Has a designated caregiver (eg, relative, housemate, close personal friend, or professional caregiver);

Exclusion Criteria:

1. Psychotic symptoms that are primarily attributable to delirium, substance abuse, or another general-medical condition (eg, hypothyroidism) or has been diagnosed with one or more of the following psychiatric conditions:

   1. Schizophrenia, schizoaffective disorder, or other psychotic disorder that is not related to Alzheimer's dementia;
   2. Bipolar disorder;
2. Risk for suicidal behavior during the course of their participation in the study or is considered to be an imminent danger to themselves or others, in the opinion of the investigator, and/or as assessed by C-SSRS; or the patient has had 1 or more suicide attempts within 2 years prior to Screening;
3. The patient is unable or unwilling to discontinue other drugs with known psychotropic properties or any non-psychotropic drugs with known or potentially significant central nervous system effects, as reviewed by the Sponsor or designee,
4. The patient is hospitalized or receiving skilled nursing care for any medical condition other than dementia
5. The patient is bedridden or has any significant medical condition that is unstable and would either:

   1. Place the patient at undue risk from study drug or undergoing study procedures; or
   2. Interfere with the interpretation of safety or efficacy evaluations performed during the course of the study;
6. The patient is in hospice or end-of-life care;

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
BEHAVE-AD psychosis subscale score | Week 6
  The BEHAVE-AD psychosis subscale is comprised of 7 items from the paranoid and delusional ideations domain and 5 items from the hallucinations domain. The scale is rated on a 4--point scale of severity, from 0 (not present) to 3 (present, generally with an emotional and physical component). The maximum score for the psychosis subscale is 36.

SECONDARY OUTCOMES:
CGI-S score | Week 6
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (22):
  - Clinical Site, Anaheim, California
  - Clinical Site, Costa Mesa, California
  - Clinical Site, Lafayette, California
  - Clinical Site, Los Alamitos, California
  - Clinical Site, Newport Beach, California
  - Clinical Site, Orange, California
  - Clinical Site, Bonita Springs, Florida
  - Clinical Site, Brandon, Florida
  - Clinical Site, Coral Springs, Florida
  - Clinical Site, Delray Beach, Florida
  - Clinical Site, Doral, Florida
  - Clinical Site, Homestead, Florida
  - Clinical Site, Maitland, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Sarasota, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Cypress, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Bellevue, Washington
- Bulgaria (5):
  - Clinical Site, Blagoevgrad
  - Clinical Site, Cherven Bryag
  - Clinical Site, Sofia
  - Clinical Site, Stara Zagora
  - Clinical Site, Vratsa
- Croatia (2):
  - Clinical Site_2, Zagreb
  - Clinical Site, Zagreb
- Czechia (3):
  - Clinical Site, Brno
  - Clinical Site, Hradec Králové
  - Clinical Site, Prague
- Poland (2):
  - Clinical Site, Bydgoszcz
  - Clinical Site, Ścinawa
- Romania (3):
  - Clinical Site, Bucharest
  - Clinical Site, Galati
  - Clinical Site, Sibiu
- Serbia (5):
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
  - Clinical Site, Niš
  - Clinical Site, Novi Kneževac
- Slovakia (5):
  - Clinical Site, Banská Bystrica
  - Clinical Site, Bratislava
  - Clinical Site, Košice
  - Clinical Site, Krompachy
  - Clinical Site, Vranov nad Topľou
- Spain (4):
  - Clinical Site, Albacete
  - Clinical Site, Madrid
  - Clinical Site, Zamora
  - Clinical Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No